CLINICAL TRIAL: NCT02378922
Title: Autologous Transplantation and Stem Cell-Based Gene Therapy With LVsh5/C46 (CAL-1), a Dual Anti-HIV Lentiviral Vector, for the Treatment of HIV-Associated Lymphoma
Brief Title: Gene-Modified HIV-Protected Stem Cell Transplant in Treating Patients With HIV-Associated Lymphoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively closed prior to subject enrollment
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9183; NCI-2015-00149 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9183 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: AIDS-Related Hodgkin Lymphoma; AIDS-Related Non-Hodgkin Lymphoma; HIV Infection; Recurrent Hodgkin Lymphoma; Recurrent Non-Hodgkin Lymphoma
MeSH Terms: conditions — HIV Infections; Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Transplantation Conditioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (gene-modified stem cells) (Experimental): CONDITIONING: Patients undergo high-dose chemotherapy or chemoradiotherapy according to institutional guidelines.
  STEM CELL INFUSION: Patients undergo hematopoietic stem cell transplant on day 0.
  Note: Patients continue to receive HAART throughout treatment, with a 7-day break for apheresis. Patients may be eligible for a structured treatment interruption of up to 12 weeks after autologous hematopoietic stem cell transplant with gene-modified cells.
  Interventions: Biological: Gene-Modified HIV-Protected Hematopoietic Stem Cells; Other: Laboratory Biomarker Analysis; Other: Transplant Conditioning

INTERVENTIONS:
Biological: Gene-Modified HIV-Protected Hematopoietic Stem Cells — Receive LVsh5/C46 (Cal-1) transduced CD34+ HSPC IV
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Transplant Conditioning — Undergo high-dose chemotherapy or chemoradiotherapy
  Other Names: conditioning regimen

SUMMARY:
This clinical trial studies gene-modified, human immunodeficiency virus (HIV)-protected stem cell transplant in treating patients with HIV-associated lymphoma. Stem cells, or cells which help form blood, are collected from the patient and stored. They are treated in the laboratory to help protect the immune system from HIV. Chemotherapy is given before transplant to kill lymphoma cells and to make room for new stem cells to grow. Patients then receive the stem cells that were collected from them before chemotherapy and have been genetically modified to replace the stem cells killed by the chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and feasibility of infusing gene-modified, HIV-protected hematopoietic stem/progenitor cells (HSPC) after high-dose chemotherapy for treatment of acquired immune deficiency syndrome (AIDS)-related lymphoma.

II. To observe the change in gene-modified cell levels before and after antiviral treatment interruption.

SECONDARY OBJECTIVES:

I. To evaluate the molecular and clonal composition of gene-modified cells after hematopoietic cell transplant (HCT).

II. To describe time to disease progression, progression-free survival, treatment-related mortality, time to neutrophil and platelet recovery, and incidence of infections.

TERTIARY OBJECTIVES:

I. To evaluate the effect of procedure on HIV-specific immune reconstitution.

II. To observe the effect of HIV infection on the presence of gene-marked cells as determined by deoxyribonucleic (DNA) polymerase chain reaction (PCR).

OUTLINE:

CONDITIONING: Patients undergo high-dose chemotherapy or chemoradiotherapy according to institutional guidelines.

STEM CELL INFUSION: Patients undergo hematopoietic stem cell transplant with LVsh5/C46 (Cal-1) transduced autologous CD34+ hematopoietic stem/progenitor cells (HSPC) on day 0.

Note: Patients continue to receive highly active antiretroviral therapy (HAART) throughout treatment, with a 7-day break for apheresis. Patients may be eligible for a structured treatment interruption of up to 12 weeks after autologous hematopoietic stem cell transplant with gene-modified cells.

After completion of study treatment, patients are followed up periodically for 2 years, every 6 months for 3 years, and then annually for 15 years post-HCT.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 seropositive
* Stable, continuous antiretroviral treatment for at least three months before enrollment, defined as a multi-drug regimen (excluding azidothymidine [AZT])
* HIV plasma viral load < 50 copies/ml
* Non-Hodgkin or Hodgkin lymphoma without active central nervous system (CNS) involvement associated with poor prognosis with medical therapy alone or for which autologous peripheral blood stem cell (PBSC) transplant is indicated:

  * Hodgkin's lymphoma beyond first remission or first partial remission or induction failure with subsequent response to salvage therapy
  * Non-Hodgkin's lymphoma beyond first remission or first partial remission or induction failure with subsequent response to salvage therapy
  * Chemotherapy responsive disease
* Karnofsky performance score >= 70%
* Subjects must agree to use effective contraception from enrollment through completion of the study
* Female subjects: if of child bearing potential, must have negative serum or urine pregnancy test within 7 days of enrollment
* Subjects must be on a prophylactic regimen for pneumocystis carinii pneumonia, or agree to begin such treatment, if CD4+ cell counts are observed to be =< 200/ul in peripheral blood
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Renal disease: serum creatinine > 2 times upper limit of normal
* Liver disease: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 3 times the upper limits of normal, unless determined to be a result of the primary hematologic malignancy
* Serum bilirubin greater than 3 times the upper limit of normal, unless attributed to Gilbert's syndrome
* Pulmonary disease: forced vital capacity (FVC) < 60% predicted
* Pulmonary disease: forced expiratory volume in 1 second (FEV1) < 60% predicted
* Pulmonary disease: diffusion capacity of the lung for carbon monoxide (DLCO) parameters < 60% predicted (corrected for hemoglobin)
* Cardiac insufficiency: left ventricular ejection fraction (LVEF) < 50% or coronary artery disease requiring treatment
* Active infection requiring systemic antibiotic therapy with antibacterial, antifungal, or antiviral agents (excluding HIV)
* Hepatitis B surface antigen positive
* Hepatitis C virus (HCV) antibody positive and detectable HCV quantitative ribonucleic acid (RNA) with clinical evidence of cirrhosis
* Requiring active treatment for Toxoplasma gondii
* Planned radiation therapy after transplant
* Malignancy other than lymphoma, unless (1) in complete remission and more than 5 years from last treatment, or (2) cervical/anal squamous cell carcinoma in situ or (3) superficial basal cell and squamous cell cancers of the skin
* History of HIV-associated encephalopathy; dementia of any kind; seizures in the past 12 months; any perceived inability to directly provide informed consent (Note: Consent may not be obtained by means of a legal guardian)
* A medical history of noncompliance with HAART or medical therapy
* Any concurrent or past medical condition that, in the opinion of the Investigator, would exclude the subject from participation or any psychosocial conditions that would hinder study compliance or follow-up, at the discretion of the Investigator
* Receipt of a vaccine for HIV-1 or any prior gene modified cell product, at any time
* Known hypersensitivity to any of the products used in the trial-G-CSF (Neupogen), plerixafor, or any planned components of conditioning regimens
* Pregnant or nursing women

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06-22 (Actual); Primary Completion 2019-06-15 (Estimated); Study Completion 2019-06-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility of collection of >= 2.1 x 10^6 CD34+ cells/kg for backup cryopreservation and collection of an additional >= 2.5 x 10^6 CD34+ cells/kg for genetic modification | Up to 15 years
Feasibility of genetic modification, defined as evidence for gene modified CD34+ cells in the infusion product | Up to 15 years
Feasibility of infusion of gene-modified cells, defined as engraftment of >= 1% gene-modified cells at the time of hematopoietic recovery from conditioning (absolute neutrophil count >= 500/mcL, platelets >= 100,000/mcL for three consecutive evaluations) | Up to 15 years
Feasibility of stem cell infusion (STI), defined as the ability to achieve engraftment level and maintain CD4 counts and plasma viremia at levels required for STI eligibility | Up to 15 years
Incidence of >= grade 3 toxicity related to the infusion of gene-modified cells, defined by Common Terminology Criteria for Adverse Events version 4.0 | Up to 15 years
Incidence of confirmed insertional mutagenesis | Up to 15 years
Incidence of development of confirmed replication competent lentivirus | Up to 15 years
Integration sites of vector sequences in peripheral blood mononuclear cells | Up to 15 years
  Characterized if clinical symptoms suggest clonal expansion of the HSPC or if molecular assays result in clonal expansion in > 20% of gene-marked cells.

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Peter Kiem, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No